CLINICAL TRIAL: NCT01608152
Title: Using Game Mechanics to Improve Outcomes Among Stem Cell Transplant Survivors
Brief Title: Development of a Video Game for the Improvement of Outcomes in Stem Cell Transplant Survivors
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2012-0362; NCI-2020-00573 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0362 (Other: M D Anderson Cancer Center); R41CA168107 (NIH)
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia; Lymphoma; Game mechanics; Stem cell transplant survivors; Hematopoietic stem cell transplantation; HSCT; Internet-based; Interactive and personalized intervention; Questionnaires; Focus groups; Interviews
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I (focus group): Patients attend a focus group for up to 1.5 hours and provide feedback on design elements, specific desirable features, and preferences for the initial prototype.
  Interventions: Behavioral: Focus Group
- Group II (access to the game): Patients have access to the game for 3 weeks and then provide feedback on problems or questions regarding the use of the prototype.
  Interventions: Other: Internet-Based Intervention; Behavioral: Interview

INTERVENTIONS:
Behavioral: Focus Group — Attend a focus group
  Groups: Group I (focus group)
Other: Internet-Based Intervention — Have access to the game
  Groups: Group II (access to the game)
Behavioral: Interview — 1 week after the 3-week period ends, interview conducted over the phone or at a clinic visit.
  Groups: Group II (access to the game)

SUMMARY:
This trial collects feedback from patients to develop a video game in improving the outcomes in stem cell transplant survivors. A video game may help to improve health behaviors for leukemia or lymphoma patients after stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop a prototype intervention electronic game that implements a baseline testable feature set, including features for social networking within a virtual game space, managing an intermittent mediated reward cycle, goal setting and tracking, and collaborative problem solving.

II. Evaluate the technical merit, feasibility, user perception and acceptance of the prototype system with adolescents and young adults (AYAs) allogeneic hematopoietic stem cell transplantation (HSCTs) patients in recovery.

III. Based on the results of the prototype evaluation, enhance and complete development of the Stempowerment on-line intervention.

IV. This is a single arm study with no comparison group; therefore, the purpose is to evaluate the impact of the Stempowerment intervention on

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients attend a focus group for up to 1.5 hours and provide feedback on design elements, specific desirable features, and preferences for the initial prototype.

GROUP II: Patients have access to the game for 3 weeks and then provide feedback on problems or questions regarding the use of the prototype.

ELIGIBILITY:
Inclusion Criteria:

Phase I

The target population for this study will consist of:

1. Individuals ages 15-29
2. Able to read and speak English
3. Diagnosis of leukemia or lymphoma
4. First time allogeneic SCT recipient

Phase II

The target population for this study will consist of:

1. Individuals ages 18-39 (in phase I, we recruited only individuals age 15-29. For phase II, we will recruit young adults, and will expand the eligible age range up to 39 years. This expansion in age eligibility to 39 years is consistent with the National Cancer Institute definition of adolescents and young adults with cancer, and is consistent with the age range of patients seen at MD Anderson in the Adolescent and Young Adult Center.
2. Able to read and speak English
3. Diagnosis of leukemia or lymphoma (including Myelodysplastic Syndrome - MDS) or lymphoma
4. HSCT recipient

Exclusion Criteria:

Phase I

The target population will be excluded if:

1. They do not speak English
2. They have vision problems
3. They have cognitive problems
4. They have psychological difficulties

Phase II

The target population will be excluded if:

1. They do not speak English
2. They have vision problems that would preclude them from viewing a computer screen.
3. They have an intellectual deficiency that would prevent the potential participant from understanding information delivered on the computer platform or as defined by the DSM-V Diagnostic and Statistical Manual of Mental Disorders that would prevent them from understanding information delivered on the computer platform.

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with leukemia or lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of electronic game intervention | 4 weeks
  Primary feasibility benchmark based on responses to questions regarding users' perceptions of the technology. If 75% of respondents have a mean score reflecting positive responses (e.g., strongly agree or agree) to each of the 7 constructs related to users' perceptions, as described above, then feasibility benchmark met. Responses to open-ended questions analyzed qualitatively using Atlas.ti software. Responses to individual questions evaluated to look for common themes, and findings used to inform future development of the prototype.

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Peterson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org